CLINICAL TRIAL: NCT02187289
Title: Night-time Compression for Breast Cancer Related Lymphedema (LYNC): A Randomized Controlled Efficacy Trial
Brief Title: Studying if Adding Night Compression to Standard Care Will Have Improved Control of Lymphedema in Breast Cancer Subjects
Acronym: LYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA CC-14-0066
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer; Lymphedema
Keywords: NCSG; Compression bandages; devices; Night time compression; Breast cancer treatment side effects; Compression therapy; Reid Sleeve; Comprefit; Medassist; Tribute; Comprilan
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard care (Active Comparator): Weeks 1-12, Standard Care only (Compression Sleeve, daytime wear)
  Interventions: Device: Compression Sleeve, daytime wear
- Standard Care plus Night-time Compression Bandages (Experimental): Weeks 1 - 12, Daytime compression sleeve plus night-time compression by self-administered or assisted multi-layered Compression Bandages.
  Interventions: Device: Night-time compression bandages; Device: Compression Sleeve, daytime wear
- Standard Care Plus Night-time Compression System Garment (Experimental): Weeks 1 - 12, Standard care (day-time sleeve) plus night-time use of a custom-made Night-time Compression System Garment
  Interventions: Device: Compression Sleeve, daytime wear; Device: Night-time Compression custom-made garment

INTERVENTIONS:
Device: Night-time compression bandages — Daytime compression sleeve plus night-time compression by self-administered or assisted multi-layered compression bandages.
  Arms: Standard Care plus Night-time Compression Bandages
Device: Compression Sleeve, daytime wear
Device: Night-time Compression custom-made garment — Standard Care plus night-time compression by a custom-made night time compression system garment.
  Arms: Standard Care Plus Night-time Compression System Garment

SUMMARY:
Lymphedema (significant arm swelling on the surgical side) is one of the most common complications following treatment for breast cancer. The impact of lymphedema is profound, resulting in negative self image, increased anxiety and poorer quality of life. In time, lymphedema can result in recurrent infections in the arm, functional impairment and pain. Approximately 21% of women who undergo breast cancer treatment develop lymphedema. Unfortunately this is a life-time condition which tends to worsen over time. Currently, treatment consists of intensive physiotherapy, meant to reduce the arm volume followed by the wearing of compression sleeves during the day for maintenance. This study hopes to show that the addition of night-time compression creates a measurable reduction in arm volume and that adding night-time compression to the standard care (daytime compression only) will produce improvements in quality of life for breast cancer survivors.

DETAILED DESCRIPTION:
Lymphedema is a lifetime condition which tends to worsen over time, affecting roughly 21% of of treated breast cancer patients. An initial intensive rehabilitative treatment is usually prescribed to reduce the lymphedema, followed by a maintenance program using compression sleeves (Standard Care). However, compression sleeves are prescribed for daytime use only due to the potential tourniquet effect of the sleeve rolling up or bunching during the night.

Compression Bandages (short stretch, low elasticity) can be used at night but proper application takes 20-30 minutes, require skill to apply properly and are costly. Various types of night-compression system garments (NCSGs) have been designed as alternatives to Compression Bandages (CB).

The objectives of this study are to determine:

1. Whether the addition of night-time compression (using CB or NCSG) to standard care (daytime compression only) improves control of arm lymphedema.
2. Whether the use of NCSGs result in better outcomes in quality of life, sleep, treatment compliance and patient independence than use of Compression Bandages.

The hypotheses are that:

1. Standard care plus the addition of NCSG will provide statistically significant improvement in management of arm lymphedema volume compared to standard care alone at 12 weeks.
2. Standard care plus the addition of Compression Bandages will provide statistically significant improved management of arm lymphedema volume compared to standard care alone at 12 weeks.
3. Standard care plus the addition of NCSG will provide statistically significant benefit in quality of life, sleep and self-efficacy over standard care plus Compression Bandaging at 12 weeks.

Group 1: Standard care weeks 1 - 12 Group 2: Standard care plus night-time Compression Bandaging weeks 1 - 12 Group 3: Standard care plus night-time use of NCSG weeks 1 - 12

All three groups will adopt NCSG use after the 12 week assessments have been done (weeks 13 - 24).

Sample size = 40 participants per group, for a total of 120 patients at three sites.

Participants will be randomized in a 1:1:1 ratio to Standard, CB or NCSG using a secure central randomization service administered by the Clinical Trials Unit of the Cross Cancer Institute. Women enrolled in the study will be stratified by accruing site and by lymphedema severity (i.e. mild versus moderate lymphedema as per the classification criteria of the International Society of Lymphology).

Arm volume (by Perometer) and arm fluid (by Bioimpedance analysis) will be measured and compared to that of the unaffected arm. BIA measures the impedance of flow from a low alternating electrical current that is applied to the body through a skin electrode. BIA records impedance values for each limb and provides an index that correlates with quantitative measurements of volume increase in limb size seen in the arm with lymphedema. This measurement will provide information on extracellular fluid changes that complements the data on arm lymphedema volume. An Independent Assessor unaware of treatment allocation (blinded) will perform the measurements of arm volume using the perometer, bioimpedance analysis, and body weight at baseline, 6, 12, 18 and 24 weeks. The duration of the primary intervention will be 12 weeks. Following the 12-week intervention period, participants in the CB and standard care groups will be measured for a NCSG.

The follow-up period after the intervention (weeks 13 to 24) will follow a longitudinal observational design and provide an opportunity to examine factors related to long-term adherence to night-time compression. Lymphedema specific questionnaires and subject diary will be completed at 6, 12, 18 and 24 weeks to assess subject's Quality of Life, sleep disturbance, self-efficacy and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer with mild to moderate lymphedema (minimum of 200 mls or 10% and maximum 40% increase in arm volume over the unaffected arm.)
* Completion of all primary and adjuvant cancer treatments (with exception of endocrine treatment) 1 month prior to randomization.
* In or entering upon the maintenance phase of lymphedema treatment.
* Have properly fitted day-time compression sleeve and agree to wear sleeve for the 12 hour per day standard of care period
* No current use of night-time compression (one month wash-out period before trial entry)

Exclusion Criteria:

* Clinical or radiological evidence of active disease, either local or metastatic
* History or clinical diagnosis of bilateral arm lymphedema
* Anyone for whom compression is contraindicated, such as those with untreated infections, skin irritations/rash, or thrombosis of the affected arm
* Serious non-malignant disease or any disorder/circumstance (psychiatric or addictive disorder) which would preclude consent/adherence to the protocol
* Unable to comply with the protocol, measurement and follow-up schedule due to factors such as vacation during the study period

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2017-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Arm volume. Lymphedema will be objectively measured using the Perometer (Pero-systems, Wipputal, Germany) | 12 weeks

SECONDARY OUTCOMES:
Arm fluid. Bioimpedance analysis (BIA) will be used to assess extracellular fluid status within the arm | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, PhD, Principal Investigator — Cross Cancer Institute
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Mount St. Joseph Hospital/Holy Family (MSJ/HF), Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available via the University of Alberta's DATAVERSE platform.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available starting 6 months after publication with no defined end date.
Access Criteria: Guest book - visitors can request the data from corresponding author.
URL: https://dataverse.library.ualberta.ca/

REFERENCES:
- [Derived] McNeely ML, Dolgoy ND, Rafn BS, Ghosh S, Ospina PA, Al Onazi MM, Radke L, Shular M, Kuusk U, Webster M, Campbell KL, Mackey JR. Nighttime compression supports improved self-management of breast cancer-related lymphedema: A multicenter randomized controlled trial. Cancer. 2022 Feb 1;128(3):587-596. doi: 10.1002/cncr.33943. Epub 2021 Oct 6. PMID 34614195
- [Derived] McNeely ML, Campbell KL, Webster M, Kuusk U, Tracey K, Mackey J. Efficacy of night-time compression for breast cancer related lymphedema (LYNC): protocol for a multi-centre, randomized controlled efficacy trial. BMC Cancer. 2016 Aug 4;16:601. doi: 10.1186/s12885-016-2648-8. PMID 27491361